CLINICAL TRIAL: NCT03805451
Title: Life Steps for PrEP for Youth
Acronym: LSPY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fenway Community Health (Other)
Collaborators: Massachusetts General Hospital (Other); University of North Carolina (Other); Emory University (Other); Brown University (Other); Cook County Hospital (Other)
Responsible Party: Principal Investigator, Kenneth H. Mayer, MD, Medical Research Director, Co-Chair TFI, Fenway Community Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ATN 158
Record Dates: First submitted 2018-05-08; First posted 2019-01-15 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: HIV; Pre-exposure Prophylaxis; Medication Adherence
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Life Steps for PrEP for Youth (Experimental): Life Steps for PrEP for Youth was derived from our prior PrEP work supported by the National Institute of Mental Health and will be tailored for YMSM/TWSM based on the findings from 20 qualitative interviews with YMSM and TWSM and 10 qualitative interviews with key informants. It will likely consist of four weekly sessions at the time of PrEP initiation and two booster sessions, which occur two and three months after PrEP initiation. Overall, the core components of the intervention will focus on medication adherence, sexual behavior, and problem solving barriers to adherence, using motivational interviewing when needed.
  Interventions: Behavioral: Life Steps for PrEP for Youth
- Standard of Care (No Intervention): After being prescribed PrEP, participants will receive standard-of-care adherence support for PrEP. They will have blood collected for medication adherence measures and will complete computer assisted behavioral surveys during study visits. Participants in this arm will also be followed for 6 months.

INTERVENTIONS:
Behavioral: Life Steps for PrEP for Youth — Life-Steps is a modular adherence intervention based on principles of cognitive-behavioral therapy (CBT), that allows for recipients of the intervention to focus on the greatest challenges that they perceive in maintaining optimal adherence to pre-exposure prophylaxis.
  Arms: Life Steps for PrEP for Youth

SUMMARY:
This is a formative study, designed to provide information required to tailor Life-Steps for Pre-Exposure Prophylaxis (PrEP), an evidence-based cognitive behavioral adherence intervention, to enhance PrEP uptake and adherence in high risk young men who have sex with men (YMSM) and young transgender women who have sex with men (YTWSM).

Life-Steps for Pre-exposure prophylaxis (PrEP) is a manualized modular adherence intervention based on principles of cognitive-behavioral therapy (CBT), that allows for recipients of the intervention to focus on the greatest challenges that they perceive in maintaining optimal adherence to PrEP.

DETAILED DESCRIPTION:
Aim 1:

To adapt Life-Steps for Pre-Exposure Prophylaxis (PrEP) to be culturally relevant and appropriate for at-risk young men who have sex with men (YMSM) and transgender women who have sex with men (TWSM). The investigators will conduct in-depth qualitative interviews with up to 20 HIV-uninfected, at risk YMSM/TWSM at Fenway Health, an Adolescent Trials Network (ATN) clinical center. The investigators will also conduct in-depth, individual qualitative interviews with up to 10 key informants, including PrEP providers and staff at community-based organizations that work with YMSM/TWSM. Through these interviews, perceived facilitators and barriers to initiating and adhering to PrEP will be identified, and potential strategies to optimize adherence to PrEP for YMSM/TWSM. The investigators will explore youth perspectives on the use of nurses to deliver health messages and weekly text messages. YMSM/TWSM will be recruited at various points in the PrEP continuum of care, including those have opted not to initiate PrEP despite recommendations from clinicians, those who are using PrEP who report high levels of adherence and those who report adherence challenges through clinician referrals and direct recruitment in clinic waiting areas. Interviews will last approximately 60 minutes and will be digitally-recorded. Recordings will be transcribed and analyzed rapidly to inform the design of the youth-tailored Life-Steps for PrEP for YMSM/TWSM that we will test in Aim 2.

Aim 2:

To conduct a 2-arm pilot randomized control trial (RCT) to assess feasibility and acceptability of the Life-Steps for PrEP for youth intervention and preliminary efficacy of the intervention to improve PrEP adherence and retention in PrEP care compared to the standard of PrEP care at three different clinical sites. Investigators will enroll 50 YMSM/TWSM in the RCT (randomized 1:1 to the 2 arms) across the 3 sites. The primary efficacy outcomes will be PrEP adherence-as measured by dried blood spot testing -and retention in PrEP care-as measured by attendance at quarterly clinic appointments-at 3 and 6 months post baseline. Secondary outcomes include changes in sexual behaviors, retention in prevention services, and acceptability of the interventions which will be assessed at each major visit. Investigators will also conduct a brief, 15-minute semi-structured exit interview with participants in the Life-Steps for PrEP for youth intervention arm to provide an opportunity for more in-depth (open-ended) feedback on intervention satisfaction and acceptability. These data will be used to finalize the intervention manual to enhance participant acceptability.

ELIGIBILITY:
Inclusion Criteria:

* age 16-24
* HIV-uninfected by self-report
* Assigned male sex at birth
* self-identify as a man who has sex with men or a trans woman who has sex with men
* able to understand English

Self-reported HIV risk is defined as meeting at least one of the following criteria:

* At least one episode of unprotected anal intercourse with an HIV-positive partner with a penis or a partner with a penis of unknown HIV status during the last 6 months;
* Anal intercourse with 3 or more partners with a penis during the last 6 months;
* Exchange of money, gifts, shelter or drugs for anal sex with a partner with a penis during the last 6 months;
* Sex with a partner with a penis and has had an STI(sexually transmitted infection) during the last 6 months;
* Sexual partner of an HIV-positive person with a penis with whom condoms were not consistently used in the last 6 months; or
* At least one episode of anal intercourse where the condom broke or slipped off during the last 6 months

Exclusion Criteria:

* Currently enrolled in another PrEP adherence study*
* Prior enrollment in an HIV vaccine trial with receipt of experimental vaccine product.*
* Enrollment in earlier phase of Life Steps for PrEP for Youth*
* Unable to give informed consent/assent due to severe mental or physical illness/substance intoxication at baseline visit
* Has severe cognitive limitation that would limit their ability to comprehend the informed consent or assent
* Presence of an active (i.e. untreated) and interfering psychiatric disorder (e.g., bipolar disorder, schizophrenia, substance abuse)

Ages: 16 Years to 24 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2019-09-27 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
Pre-Exposure Prophylaxis (PrEP) Adherence at 3 months post PrEP initiation | Blood sample collected at 3 month visit post baseline
  Measured by dried blood spot (DBS) testing of tenofovir diphosphate (TFV-DP) and emtricitabine triphosphate (FTC-TP)
Pre-Exposure Prophylaxis (PrEP) Adherence at 6 months post PrEP initiation | blood sample collected at 6 month visit post baseline
  Measured by dried blood spot (DBS) testing of tenofovir diphosphate (TFV-DP) and emtricitabine triphosphate (FTC-TP)

SECONDARY OUTCOMES:
Retention in Pre-Exposure Prophylaxis (PrEP) care and prevention services | Records will be abstracted at the end of the study period for each participant to determine if they attended a clinic appointment at 3 and 6 months post baseline
  Attendance at quarterly clinic appointments obtained through medical record abstraction
LifeSteps for PrEP for Youth Intervention Acceptability | Measured at each study visit (3 and 6 months post baseline)
  To measure acceptability, participants will be asked to self-report the degree to which they find the intervention appropriate and useful using Likert-type agreement scales.
LifeSteps for PrEP for Youth Intervention Satisfaction | Measured at each study visit (3 and 6 months post baseline)
  Satisfaction will be measured with the Client Satisfaction Questionnaire (CSQ-8). The CSQ-8 is an 8-item, easily scored and administered measurement designed to measure client satisfaction with services.
  The CSQ-8 has been extensively studied, and while it is not necessarily a measure of a client's perceptions of gain from treatment, or outcome, it does elicit the client's perspective on the value of services received. The CSQ-8 seems to operate about the same across all ethnic groups.
  The CSQ-8 is scored by summing the item scores to produce a range of 8 to 32, with high scores indicating greater satisfaction.
  Larsen, D.L., Attkisson, C.C., Hargreaves, W.A., and Nguyen, T.D. (1979). Assessment of client/patient satisfaction: Development of a general scale, Evaluation and Program Planning, 2, 197-207. Instrument reproduced with permission of C. Clifford Attkisson. Attkisson, C. C., & Greenfield, T. K. (1994). Client Satisfaction Questionnaire-8 and Service Satisfaction Scale-30.

OTHER OUTCOMES:
Adapt Life-Steps for PrEP to be appropriate for at-risk young men who have sex with men (YMSM) and young transgender women who have sex with men (YTWSM) | one time qualitative interviews will be conducted
  Study Investigators will conduct qualitative interviews with up to 20 HIV-uninfected YMSM/TWSM at Fenway Health and with up to 10 key informants, including PrEP providers and staff at community-based organizations that work with YMSM/TWSM. Interviews will be transcribed and analyzed using content analysis to identify changes that should be made to the Life-Steps intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Ken A Mayer, MD, Principal Investigator — The Fenway Institute; Christina Psaros, Ph.D., Principal Investigator — Harvard Medical School and Massachusetts General Hospital
Locations (3):
- United States (3):
  - PRISM Health, Atlanta, Georgia
  - Core Center, Chicago, Illinois
  - Fenway Health, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No